CLINICAL TRIAL: NCT03103113
Title: Division of Infertility, Lee Women's Hospital, Taichung, Taiwan
Brief Title: The Evolution of Relationship Between Results of Peripheral Blood Test and Outcomes of in Vitro Fertilization
Status: Completed | Type: Observational
Sponsor: Yeh (Other)
Responsible Party: Sponsor-Investigator, Yeh, institutional review board, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Other Study IDs: CS12033
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Infertility, Female; Immune Tolerance
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The purpose of this study was to assess the relationship between infertility blood test results and outcomes of pregnancy and alive birth of women who underwent with or without intravenous immunoglobulin (IVIG) before in vitro fertilization.

DETAILED DESCRIPTION:
Study Design (Brief Description)

1. Inclusion criteria Patients had underwent infertility blood test or treatment in Lee's women hospital
2. Exclusion criteria No
3. Endpoint

1. Values of blood test (PTT, IDM, ANA, Lupus, protein-s) 2. Embryo quality 3. Results of intravenous immunoglobulin (IVIG) treatment (pregnancy or not) 4. Alive birth rate

4. Withdraw criteria and rescue medication No 5. Sample Size and Study Duration Sample Size: total 500 women who underwent IVF treatments and tests from Jan. 2007 to Dec. 2010.

Study Duration: from date of IRB agreement to Dec. 2012 6. Please specify objectives of study when collecting extra specimen from participants No more need to collect extra specimen from participants in this study 7. Expected Endpoints of Treatment No 8. Others No

ELIGIBILITY:
Inclusion Criteria:

* Patients had underwent both infertility blood test and IVF treatment in Lee's women hospital

Exclusion Criteria:

* No

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients had underwent infertility blood test and in vitro fertilization treatment in Lee's women hospital
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
implantation rate | 6-8 weaks after last menstrual
  sac and heart bit can be detected after embryo transfer

SECONDARY OUTCOMES:
live birth rate | live birth after pregnant
  live birth after IVF treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maw Sheng Lee, Study Chair — Lee's Women Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared after manuscription publication